CLINICAL TRIAL: NCT04620291
Title: A Phase I, Open-Label, Multi-Dose Study for Evaluation of the Safety, Pharmacokinetics, and Antiviral Activity of UB-421 Subcutaneous Formulation in HIV Infected Adults
Brief Title: Study for Evaluation of the Safety, Pharmacokinetics, and Antiviral Activity of UB-421 Subcutaneous Formulation in HIV Infected Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A127-HIV
Record Dates: First submitted 2020-10-28; First posted 2020-11-06 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A (Experimental): 250 mg UB-421 SC: ART-treated subjects
  Interventions: Biological: UB-421 SC
- Cohort B (Experimental): 500 mg UB-421 SC: ART-treated subjects
  Interventions: Biological: UB-421 SC
- Cohort C (Experimental): 700 mg UB-421 SC: ART-treated subjects
  Interventions: Biological: UB-421 SC
- Cohort D (Experimental): 500 mg UB-421 SC: Treatment naive subjects
  Interventions: Biological: UB-421 SC
- Cohort E (Experimental): 700 mg UB-421 SC: Treatment naive subjects
  Interventions: Biological: UB-421 SC

INTERVENTIONS:
Biological: UB-421 SC — The UB-421 SC (dB4C7C22-6 mAb) will be supplied at a concentration of 125 mg/mL after reconstitution. Subjects will receive weekly UB-421 SC injections during the 4-week Treatment Period.
  Other Names: Humanized dB4C7C22-6 monoclonal antibody

SUMMARY:
UB-421 subcutaneous formulation (UB-421 SC) is developed to provide HIV infected patients a more convenient drug delivery method. UB-421 SC injection, with significantly less injection time than IV infusions and with opportunity of self-administration or administered in general medical setting (in addition to HIV-specific clinic), can provide patient a more convenient option.

This UB-421 SC phase I study will be conducted to investigate short-term safety, pharmacokinetics and anti-viral activity of UB-421 SC at three dose levels in ART-treated aviremic subjects and treatment naive HIV-infected subjects. The current UB-421 SC formulation (125 mg/ml) is at least 10-fold more concentrated than UB-421 IV (10 mg/ml). The highly concentrated formulation makes weekly UB-421 subcutaneous injections feasible. This study will form the basis of UB-421 SC in combination with antiretroviral agents (ARV) for treating HIV infected viremic patients in the future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

ART-treated aviremic subjects who meet all inclusion criteria (A~C and 1~5) will be eligible for Part A: A. Documentation of continuous ART treatment with suppression of plasma viral level below the limit of detection for ≥1 years. Individuals with "blips" (i.e., detectable viral levels on ART) prior to the Screening Visit (SV) may be included provided they satisfy the following criteria:

1. The blips are <400 copies/mL, and
2. Succeeding viral levels return to levels below the limit of detection on subsequent testing B. Tolerated the baseline ART regimen (without major toxicity) and are expected to continue in the trial period (since SV till EOS) the same ART regimen. The change in brand or formulation but not in the 3 ARV types (eg, from 3 tablets to 1 single tablet containing the same 3 ARV drugs, or from immediate-release to extended-release tablet per day, or other similar change are allowed) are considered the same ART regimen; C. Viral load should below 50 RNA copies/mL at the SV; ART-naïve viremic subjects who meet all inclusion criteria (D~F and 1~5) will be eligible for

Part B:

D. HIV-1 viral load >200 copies/mL at the SV; E. HIV antiretroviral therapy (ART)-naïve i.e., subjects who receive no prior or current ART.

However, subjects who have previously received pre- or post-exposure prophylaxis but eventually confirmed HIV-1 seropositive can be enrolled; F. Asymptomatic (generalized lymphadenopathy can be included), defined as subjects without stage 3 defining opportunistic illnesses according to revised Surveillance Case Definition for HIV Infection published in 2014, which was determined by the Investigator based on the medical history, physical examination, ECG, and laboratory evaluations;

Inclusion criteria for both Part A and B:

1. HIV-1 seropositive, with documented HIV-1 infection by official, signed, written history (e.g.

   laboratory report);
2. Male and female, age 18 years or older;
3. CD4+ (D1) T cell count > 350 cells/mm3 at the SV;
4. Male subjects and female subjects of childbearing potential must agree to use the acceptable method of contraception during the course of the study (excluding women who are not of childbearing potential). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at the SV; Definitions Women NOT of childbearing potential: women who are permanently or surgically sterilized or postmenopausal. Permanent sterilization includes hysterectomy, and/or bilateral oophorectomy, and/or bilateral salpingectomy and/or tubal ligation.

   Postmenopausal women: 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. Acceptable method of birth control for WOCBP: abstinence; implant; intrauterine device; hormonal contraceptive (injectable, oral contraceptives, transdermal patches, or contraceptive rings) plus barrier method (male condom, female condom or diaphragm). Acceptable method of birth control for male subjects: abstinence; condom.
5. Subjects signed the informed consent before undergoing any study procedures.

Exclusion Criteria:

Subjects who have any of the following conditions will be excluded from both Part A and B

1. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study;
2. Subjects with acute opportunistic infection(s) or bacterial infection(s), that the delayed initiation of ART would not be allowed, as judged by the Investigator;
3. Any stage 3 defining opportunistic illnesses such as Kaposi's sarcoma according to the revised Surveillance Case Definition for HIV Infection published in 2014 within the past 12 months before the SV;
4. Serious illness requiring systemic treatment and/or hospitalization for at least 7 days prior to the SV;
5. Any previous exposure to a monoclonal antibody within 12 weeks prior to the SV;
6. Any previous hypersensitivity reaction to monoclonal antibody;
7. Have ever experienced urticaria in the previous 2 years before the SV or with ongoing dermatologic problem with rash appearance (eg. eczema, atopic dermatitis, urticaria) at the SV;
8. Any significant diseases (other than HIV-1 infection) or clinically significant findings that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy;
9. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
10. Presence of hepatitis B surface antigen (HBsAg) or HCV antibody and RNA double positive at the Screening Visit or within 12 weeks prior to the SV;
11. Serum GPT/ALT value is 2.5 times or greater than the upper limit of normal (≥ 2.5 xULN) at the Screening Visit;
12. Serum GOT/AST value is 2.5 times or greater than the upper limit of normal (≥ 2.5 xULN) at the Screening Visit;
13. Serum total bilirubin (TBIL) value is 2.5 times or greater than the upper limit of normal (≥ 2.5 xULN) at the SV;
14. Serum creatinine value is greater than 1.5 times the upper limit of normal (> 1.5 x ULN) at the SV;
15. Any vaccination within 8 weeks prior to the SV;
16. Any treatment with immunomodulators, such as interleukins, interferon, cyclosporine, systemic corticosteroid, or systemic chemotherapy within 12 weeks prior to the Screening Visit; Note: Subjects received short-term low dose oral (i.e. prednisone ≤0.5mg/kg/day f or ≤ 1 - month duration), inhaled, nasal, or topical steroids will not be excluded.)
17. Prior participation in any HIV vaccine trial;
18. Receipt of other investigational study agent within 12 weeks before the SV;
19. Life expectancy of less than 12 months;
20. Any current alcohol or illicit drug use that, in the Investigator's opinion, would interfere with the subject's ability to comply with the dosing and visit schedules and protocol evaluations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Numbers and incidence of TEAEs | 28 days
  Numbers and incidence of TEAEs that are ≥ Grade 2 and study treatment related, TEAEs (any grades) by maximum severity, TEAEs by relationship to study treatment, SAEs, TEAEs leading to death, and TEAEs leading to discontinuation of study treatment will be tabulated by dose cohort and will be summarized by system organ class and preferred term for study period (Treatment or Follow-up). The "Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events" will be used in this study for all AE severity grading, except skin abnormalities, which will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
The virologic responses during the Treatment Period | 28 days
  The proportion of subjects ever achieving HIV-1 RNA reduction > X log10 copies/mL;
PK of UB-421 SC | 28 days
  • Ctrough for each dosing interval;
PK of UB-421 SC | 28 days
  Cmax of first dosing interval;
PK of UB-421 SC | 28 days
  AUC0-inf (if applicable).

OTHER OUTCOMES:
Serum anti UB-421 antibody level | 49 days
  Serum levels of anti-UB-421 antibody